CLINICAL TRIAL: NCT06704178
Title: A Randomized Double-blind Placebo-controlled Study to Evaluate the Effects of a Dietary Supplement on Children's Health and Development Outcomes.
Brief Title: A Study to Evaluate the Effects of a Dietary Supplement on Children's Health and Development Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuBest (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 20424
Record Dates: First submitted 2024-08-07; First posted 2024-11-26 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Height; Cognitive Function; Weight Gain
Keywords: Dietary Supplement; Growth and Development
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, two-arm trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is double-blind; participants, care providers, investigators, and outcomes assessors are all masked to the allocation of intervention or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in this arm will take NuBest Tall Growth Protein Powder daily for 6 months.
  Interventions: Dietary Supplement: NuBest Tall Growth Protein Powder
- Placebo Arm (Placebo Comparator): Participants in this arm will take a placebo product daily for 6 months.
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: NuBest Tall Growth Protein Powder — NuBest Tall Growth Protein Powder includes a proprietary blend of vitamins, minerals, and probiotics designed to enhance children's health outcomes.
  Arms: Intervention Arm
Dietary Supplement: Placebo Powder — The placebo powder is designed to mimic the appearance and taste of the NuBest Tall Growth Protein Powder but does not contain the active ingredients.
  Arms: Placebo Arm

SUMMARY:
A 6-month virtual two-armed randomized double-blind placebo-controlled clinical trial. Participants will take NuBest Tall Growth Protein Powder or a placebo daily. Parents will complete questionnaires at baseline and monthly, and children will undergo cognitive assessments and height/weight measurements at specified intervals.

ELIGIBILITY:
Inclusion Criteria:

* Interested in their child trialing a dietary supplement designed to improve overall health outcomes in children including height, maintenance of a healthy weight, cognitive function, immune function, and energy levels.
* Willing to refrain from giving their child any vitamins, minerals, or herbal supplements of any kind for the duration of the study.
* Parents willing to weigh and measure the height of their child throughout the study.
* Generally healthy - do not have any uncontrolled chronic disease.

Exclusion Criteria:

* Any child with a history of endocrine disorder, heart disease, lung disease, kidney disease, digestive disease, or skeletal dysplasia.
* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Is undergoing or planning to undergo significant medical procedures in the next six months.
* A history of severe allergic reactions, including but not limited to any of the product's ingredients.
* Any child with a dairy allergy or lactose intolerance.
* Has undergone any surgeries or invasive treatments in the last six months.
* Has had any major illness in the last three months.
* Having any planned invasive medical procedures during the study period.
* Currently participating in any other clinical study.
* Unwilling to follow the study protocol.
* Any child diagnosed with attention-deficit disorder (ADD) or attention-deficit hyperactivity disorder (ADHD).
* Any child currently taking or have taken in the last 3 months any prescription medication targeting ADD or ADHD (such as Adderall, Concerta, Focalin, Evekeo, or Ritalin).
* Any child that is a 'fussy' eater or who the parent suspects may not tolerate consuming the test product daily for six months.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-02-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: Participants in this arm will take NuBest Tall Growth Protein Powder daily for 6 months (n=30).
- Placebo Arm: Participants in this arm will take a placebo product daily for 6 months (n=30).
Period: Overall Study
Arm/Group | Intervention Arm | Placebo Arm
Started | 30 | 30
Completed | 25 | 21
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Placebo Arm | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.19 (1.75) | 12.14 (2.26) | 12.64 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 20 | 12 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change Mean Percentile Score in Double Trouble
Description: The primary outcome measure will assess the improvement in cognitive function as evaluated by a cognitive test. Participants received a percentile score (1-100) on the assessment, with a higher score indicating a better response.
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 24 | 21
percent change from baseline | 168.55 (230.40) | 129.46 (332.76)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.488445, Multiple t-tests

2. Primary Outcome: IChange Mean Percentile Score in Feature Match
Description: The primary outcome measure will assess the improvement in cognitive function as evaluated by a cognitive test. Feature Match is a focus and processing task. Participants received a percentile score (1-100) on the assessment, with a higher score indicating a better response.
Time Frame: Baseline and Month 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 24 | 21
percent change from baseline | 34.60 (67.93) | 58.20 (147.20)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority — Between-group comparison; p = 0.98317, t-test, 2 sided — Between-group comparison

3. Primary Outcome: Change Mean Percentile Score in Grammatical Reasoning
Description: The primary outcome measure will assess the improvement in cognitive function as evaluated by a cognitive test. Grammatical Reasoning is a deductive reasoning task that requires quickly interpreting phrases and making logical conclusions from understanding. Participants received a percentile score (1-100) on the assessment, with a higher score indicating a better response.
Time Frame: Baseline to Month 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 24 | 21
percent change from baseline | 56.59 (130.07) | 88.39 (214.99)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.98317, t-test, 2 sided

4. Primary Outcome: Change Mean Percentile Score in Digit Span
Description: The primary outcome measure will assess the improvement in cognitive function as evaluated by a cognitive test. Digit Span requires users to focus on displayed numbers, hold them in short-term memory, and repeat them back correctly. Participants received a percentile score (1-100) on the assessment, with a higher score indicating a better response.
Time Frame: Baseline to Month 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 24 | 21
percent change from baseline | 28.02 (60.29) | 19.69 (69.38)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.919209, t-test, 2 sided

5. Primary Outcome: Change Mean Percentile Score in Token Search
Description: The primary outcome measure will assess the improvement in cognitive function as evaluated by a cognitive test. Leveraging the brain's executive functioning skills, Token Search requires participants to hold information in working memory and remain focused on completing sequential steps. Participants received a percentile score (1-100) on the assessment, with a higher score indicating a better response.
Time Frame: Baseline to Month 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 24 | 21
percent change from baseline | 6.26 (36.38) | 40.20 (145.02)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.919209, t-test, 2 sided

6. Secondary Outcome: Increase in Height
Description: Height measurement will be taken using an Ultrasonic Height Measuring Stadiometer. The increase in height will be tracked over the course of the study.
Time Frame: Baseline, Month 2, Month 4, and Month 6
Population: The number of participants analyzed at each time point reflects the available data from participants who completed assessments at that specific time point. The decreasing numbers are due to participant dropouts and missed measurements. All data were analyzed using an intention-to-treat (ITT) approach, with results reported for all participants who provided data at each respective time point.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 25
percent change from baseline
  Month 2 | 0.89 (4.01) | 1.16 (6.29)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 3.25 (4.19) | 1.67 (4.47)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 3.47 (5.68) | 3.49 (4.54)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.954882, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.246176, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.954882, t-test, 2 sided — Comparison at Month 6

7. Secondary Outcome: Changes in Weight
Description: Weight measurement will be taken using a FitBit Smart Scale. Changes in weight will be analyzed across the groups.
Time Frame: Baseline, Month 2, Month 4, and Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 25
percent change from baseline
  Month 2 | 4.67 (7.83) | 4.50 (14.92)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 5.52 (5.72) | 2.29 (6.80)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 7.53 (11.69) | 4.65 (5.71)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.483382, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.483382, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.726742, t-test, 2 sided — Comparison at Month 6

8. Secondary Outcome: Changes in Overall Health as Reported by Parents
Description: This parameter was assessed using a parent-completed questionnaire. Parents were required to rate their child's overall health in the past four weeks. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Very Poor" ," 5 = "Excellent"). An increase in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 0.45 (15.09) | 0.19 (31.04)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 1.22 (13.87) | 6.73 (34.70)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -0.51 (15.32) | 14.42 (28.39)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 3.75 (15.39) | 9.17 (27.69)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 1.32 (15.12) | 17.17 (40.45)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 3.27 (14.48) | 12.46 (31.13)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999216, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.559556, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999984, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.952545, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998367, t-test, 2 sided — Comparison at Month 6

9. Secondary Outcome: Change in Parents' Perception of the Child's Health in the Future.
Description: This parameter was assessed using a parent-completed questionnaire, with the question "I expect my child will have a very healthy life". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Never," 5 = "Always"). An increase in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 16.99 (60.80) | 3.53 (32.93)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 19.87 (62.14) | 7.33 (30.17)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 19.55 (60.73) | 9.78 (25.46)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 18.06 (67.82) | 4.86 (22.10)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 20.83 (62.55) | 8.33 (25.00)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 18.67 (61.44) | 8.33 (27.13)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999851, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999801, t-test, 2 sided
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999984, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.993223, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999567, t-test, 2 sided — Comparison at Month 6

10. Secondary Outcome: Parents' Perception of the Change in Child's Health Compared to One Month Ago.
Description: This parameter was assessed using a parent-completed questionnaire, whereby parents were asked to rate their child's overall health in the past 4 weeks. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Much worse," 5 = "Much Better"). An increase in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 12.82 (23.24) | 8.01 (36.25)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 18.27 (26.46) | 17.33 (38.56)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 20.19 (26.68) | 25.00 (27.75)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 19.44 (23.91) | 25.90 (42.88)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 12.85 (23.05) | 28.99 (30.96)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 24.00 (29.00) | 24.21 (25.40)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999851, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999838, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.991697, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999984, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.581904, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999866, t-test, 2 sided — Comparison at Month 6

11. Secondary Outcome: Change in Child's Energy Levels as Reported by Parents
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Very Poor," 5 = "Excellent"). An increase in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 9.17 (18.20) | 11.47 (51.50)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 5.83 (18.69) | 13.20 (20.34)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 11.86 (16.02) | 26.88 (47.45)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 18.75 (24.85) | 26.32 (66.60)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 15.14 (23.86) | 27.61 (65.04)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 16.53 (31.79) | 15.95 (28.48)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999835, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.962016, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.995044, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998665, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999816, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999567, t-test, 2 sided — Comparison at Month 6

12. Secondary Outcome: Changes in Limitations When Completing High-Intensity Activity
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where lower scores indicate better outcomes (e.g., 1 = "Never," 5 = "Always"). An increase in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 8.33 (43.27) | 3.85 (67.22)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 12.18 (46.80) | 0.00 (29.27)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 6.41 (46.92) | -13.77 (21.70)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 0.00 (25.54) | -7.64 (50.12)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 6.25 (49.59) | -13.04 (23.00)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -2.00 (26.93) | 0.00 (72.65)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999851, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999524, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.576782, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.772865, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.91384, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.992841, t-test, 2 sided — Comparison at Month 6

13. Secondary Outcome: Changes in Limitations When Completing Moderate-Intensity Activity
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). An increase in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 0.64 (41.76) | 8.33 (65.36)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 0.64 (41.76) | 4.67 (49.19)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -3.21 (36.52) | -9.42 (18.69)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -10.42 (20.74) | -11.11 (20.06)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | -2.08 (47.73) | -7.97 (18.03)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -10.00 (20.41) | -1.59 (50.53)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999732, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999801, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p > 0.999999, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999816, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p > 0.999999, t-test, 2 sided — Comparison at Month 6

14. Secondary Outcome: Changes in Limitations When Moving Around
Description: as for outcome 13
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 7.69 (27.17) | 14.10 (61.95)
  Month 2: number analyzed (Participants) | 26 | 23
  Month 2 | 7.69 (27.17) | 6.67 (40.82)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 3.85 (19.61) | -1.45 (6.95)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 0.00 (0.00) | 5.56 (42.47)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 8.33 (40.82) | 2.90 (22.28)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 0.00 (0.00) | 12.70 (48.85)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999851, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998326, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998665, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999816, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998846, t-test, 2 sided — Comparison at Month 6

15. Secondary Outcome: Changes in Limitations When Walking 100 Meters or Climbing a Flight of Stairs
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | -0.96 (26.91) | 6.41 (46.92)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 2.88 (33.41) | -1.33 (25.87)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -2.88 (28.57) | -1.45 (27.02)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -3.13 (29.77) | -1.39 (26.43)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 1.04 (46.90) | -4.35 (14.41)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -7.00 (19.79) | 14.29 (63.53)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999387, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p > 0.999999, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999984, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999816, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998367, t-test, 2 sided — Comparison at Month 6

16. Secondary Outcome: Change in Limitations When Bending, Lifting, or Stooping.
Description: as for outcome 15
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 5.77 (29.42) | 6.41 (54.79)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 3.85 (31.38) | 0.67 (34.52)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -3.85 (13.59) | -1.45 (27.02)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -2.08 (10.21) | 2.78 (44.69)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 6.25 (42.51) | -6.52 (17.22)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -2.00 (10.00) | 0.00 (27.39)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999975, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999801, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999984, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.960874, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999567, t-test, 2 sided — Comparison at Month 6

17. Secondary Outcome: Change in Limitations in the Kind of Schoolwork or Activities Undertaken.
Description: as for outcome 15
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 5.77 (29.42) | -0.96 (53.56)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 5.77 (29.42) | -4.00 (29.38)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 1.92 (22.27) | -5.43 (30.94)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -4.17 (14.12) | -10.42 (21.88)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 4.17 (44.03) | -9.42 (21.80)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -4.00 (13.84) | -7.14 (35.19)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.981906, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.945027, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.767795, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.996139, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.952378, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998846, t-test, 2 sided — Comparison at Month 6

18. Secondary Outcome: Change in Limitations in the Amount of Time Spent Completing Schoolwork or Activities.
Description: as for outcome 15
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 19.23 (51.14) | -5.13 (56.13)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 0.00 (24.49) | -3.00 (37.64)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 7.69 (36.58) | -9.78 (20.82)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -6.25 (16.89) | -10.76 (23.11)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 2.08 (45.39) | -9.42 (21.80)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -6.00 (16.58) | -7.14 (35.19)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.55783, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.987949, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.576782, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998665, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.989226, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999567, t-test, 2 sided — Comparison at Month 6

19. Secondary Outcome: Change in Limitations During the Completion of Schoolwork or Activities.
Description: as for outcome 15
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 5.77 (29.42) | -0.64 (65.06)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 9.62 (60.03) | -2.00 (37.37)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 3.85 (31.38) | -13.04 (26.09)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -6.25 (16.89) | -12.50 (23.70)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 2.08 (45.39) | -13.04 (26.09)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -6.00 (16.58) | -14.29 (27.02)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.795476, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.977286, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.559556, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.997753, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.952378, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.988108, t-test, 2 sided — Comparison at Month 6

20. Secondary Outcome: Change in Parents' Perception of Child's Health Compared to Other Children.
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "My child seems less healthy than other children". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | -1.92 (46.27) | 1.60 (47.61)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 2.56 (68.91) | -4.00 (32.38)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -16.67 (24.49) | 1.45 (53.16)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -12.50 (34.49) | 0.00 (46.88)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | -2.08 (45.92) | 15.22 (80.55)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 0.00 (43.83) | 8.73 (52.60)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.995367, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.974102, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998665, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999816, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999567, t-test, 2 sided — Comparison at Month 6

21. Secondary Outcome: Change in Parents' Perception of Child's Immunity
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "When something is going around my child usually catches it". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | -5.77 (12.19) | 18.59 (73.34)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | -11.86 (21.37) | 1.33 (25.76)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -8.01 (25.22) | 12.68 (54.98)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -9.72 (18.17) | 5.56 (53.26)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | -12.85 (29.69) | -3.99 (31.97)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -9.00 (31.91) | -1.98 (38.54)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.882016, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.860406, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.958944, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998816, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.989226, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999296, t-test, 2 sided — Comparison at Month 6

22. Secondary Outcome: Change in Parents' Worry About Child's Health
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "I worry more about my child's health than other parents do their children". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter.
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | 7.37 (69.77) | -9.29 (31.83)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | 12.18 (51.71) | 1.33 (56.91)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | 2.24 (55.81) | 1.45 (40.80)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | 4.86 (67.25) | -1.39 (48.94)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | 10.76 (55.30) | 2.54 (60.59)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | 1.33 (52.63) | -7.94 (57.40)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999975, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.977286, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999984, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.986557, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998367, t-test, 2 sided — Comparison at Month 6

23. Secondary Outcome: Change in Parent-reported Frequency of Child's Stomach Aches
Description: as for outcome 15
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | -4.49 (26.48) | -9.62 (33.72)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | -7.69 (28.37) | -11.00 (30.12)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -10.26 (24.98) | -7.97 (51.46)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -6.25 (31.40) | -11.11 (37.00)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | -13.19 (34.40) | -9.42 (32.50)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -19.33 (31.80) | -12.70 (35.32)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999851, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999801, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998467, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999816, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.998846, t-test, 2 sided — Comparison at Month 6

24. Secondary Outcome: Change in Parent-reported Frequency of Child's Difficulty Going to the Toilet
Description: as for outcome 15
Time Frame: Monthly from Baseline to Month 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 26 | 26
percent change from baseline
  Month 1 | -6.79 (28.89) | -7.05 (39.91)
  Month 2: number analyzed (Participants) | 26 | 25
  Month 2 | -10.19 (29.11) | -7.00 (38.32)
  Month 3: number analyzed (Participants) | 26 | 23
  Month 3 | -18.21 (22.79) | -11.96 (37.17)
  Month 4: number analyzed (Participants) | 24 | 24
  Month 4 | -21.53 (23.30) | -10.42 (33.27)
  Month 5: number analyzed (Participants) | 24 | 23
  Month 5 | -17.01 (36.98) | -15.58 (36.44)
  Month 6: number analyzed (Participants) | 25 | 21
  Month 6 | -21.00 (39.32) | -3.57 (37.69)
Statistical Analysis 1: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p > 0.999999, t-test, 2 sided — Comparison at Month 1
Statistical Analysis 2: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999779, t-test, 2 sided — Comparison at Month 2
Statistical Analysis 3: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999801, t-test, 2 sided — Comparison at Month 3
Statistical Analysis 4: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.963236, t-test, 2 sided — Comparison at Month 4
Statistical Analysis 5: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.999816, t-test, 2 sided — Comparison at Month 5
Statistical Analysis 6: Comparison: Intervention Arm vs Placebo Arm; Test type: Superiority; p = 0.737995, t-test, 2 sided — Comparison at Month 6

25. Secondary Outcome: Change Mean Percentile Score in Double Trouble - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed within the NuBest group using a child-completed cognitive assessment. Participants received a percentile score ranging from 1 to 100, with higher scores indicating better cognitive function. The overall score at each timepoint reflects performance on the cognitive test.
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentile score
  Baseline | 28 (22.46)
  Month 6 | 48.67 (27.18)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.0003, t-test, 2 sided — Within-group analysis only

26. Secondary Outcome: Change Mean Percentile Score in Feature Match - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 2
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentile score
  Baseline | 39.58 (17.86)
  Month 6 | 45.75 (15.26)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.2698, t-test, 2 sided — Within-group analysis only

27. Secondary Outcome: Change Mean Percentile Score in Grammatical Reasoning Match - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 3
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentile score
  Baseline | 47.42 (24.42)
  Month 6 | 56.54 (28.46)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.2698, t-test, 2 sided — Within-group analysis only

28. Secondary Outcome: Change Mean Percentile Score in Digit Span - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 4
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentile score
  Baseline | 42.29 (14.33)
  Month 6 | 50.88 (22.66)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.2137, t-test, 2 sided — Within-group analysis only

29. Secondary Outcome: Change Mean Percentile Score in Token Search - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 5
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
percentile score
  Baseline | 53.17 (17.20)
  Month 6 | 53.04 (14.44)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.8639, t-test, 2 sided — Within-group analysis only

30. Secondary Outcome: Change Mean Percentile Score in Double Trouble - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
percentile score
  Baseline | 33.73 (18.98)
  Month 6 | 49.62 (28.48)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.239, t-test, 2 sided — Within-group analysis only

31. Secondary Outcome: Change Mean Percentile Score in Feature Match - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 2
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
percentile score
  Baseline | 40.81 (19.49)
  Month 6 | 45.29 (22.87)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.6088, t-test, 2 sided — Within-group analysis only

32. Secondary Outcome: Change Mean Percentile Score in Grammatical Reasoning - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 3
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
percentile score
  Baseline | 47.05 (25.36)
  Month 6 | 54.33 (32.05)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.5738, t-test, 2 sided — Within-group analysis only

33. Secondary Outcome: Change Mean Percentile Score in Digit Span - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 4
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
percentile score
  Baseline | 52.57 (14.70)
  Month 6 | 57.62 (22.36)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.6088, t-test, 2 sided — Within-group analysis only

34. Secondary Outcome: Change Mean Percentile Score in Token Search - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 5
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: percentile score
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
percentile score
  Baseline | 48.62 (18.50)
  Month 6 | 55.62 (21.08)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.4942, t-test, 2 sided — Within-group analysis only

35. Secondary Outcome: Increase in Height - Nubest Group Only (Within-Group Analysis)
Description: as for outcome 6
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
inches
  Baseline | 61.69 (5.50)
  Month 2 | 62.01 (5.82)
  Month 4 | 63.33 (5.81)
  Month 6 | 63.24 (4.54)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.7419, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p = 0.0033, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p = 0.0219, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

36. Secondary Outcome: Increase in Height - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 6
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
inches
  Baseline | 60.66 (7.07)
  Month 2 | 62.41 (5.88)
  Month 4 | 62.71 (5.29)
  Month 6 | 63.05 (5.24)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.7708, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p = 0.239, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.006, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

37. Secondary Outcome: Changes in Weight - Nubest Group Only (Within-Group Analysis)
Description: Weight measurement will be taken using a FitBit Smart Scale.
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: Pounds
Groups:
- Intervention Arm: Participants in this arm will take the test product daily for 6 months (n=30).
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
Pounds
  Baseline | 121.68 (40.91)
  Month 2 | 126.38 (47.81)
  Month 4 | 124.36 (45.35)
  Month 6 | 123.82 (34.70)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.0219, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p = 0.0001, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p < 0.0001, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

38. Secondary Outcome: Changes in Weight - Placebo Group Only (Within-Group Analysis)
Description: Weight measurement will be taken using a FitBit Smart Scale.
Time Frame: Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: Pounds
Groups:
- Placebo Arm: Participants in this arm will take the placebo product daily for 6 months (n=30).
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
Pounds
  Baseline | 130.43 (50.58)
  Month 2 | 137.92 (57.12)
  Month 4 | 133.06 (48.91)
  Month 6 | 128.99 (46.47)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.0695, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p = 0.0124, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.0016, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

39. Secondary Outcome: Changes in Overall Health as Reported by Parents - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Parents were required to rate their child's overall health in the past four weeks. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Very Poor" ," 5 = "Excellent"). An increase in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the NuBest group only.
Time Frame: Monthly from Baseline to Month 6.
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 4.33 (0.70)
  Month 1 | 4.29 (0.62)
  Month 2 | 4.33 (0.64)
  Month 3 | 4.25 (0.68)
  Month 4 | 4.42 (0.50)
  Month 5 | 4.33 (0.64)
  Month 6 | 4.38 (0.58)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

40. Secondary Outcome: Change in Parents' Perception of the Child's Health in the Future - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Very Poor" ," 5 = "Excellent"). An increase in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the NuBest group only.
Time Frame: Monthly from Baseline to Month 6.
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 3.38 (0.77)
  Month 1 | 3.63 (0.49)
  Month 2 | 3.71 (0.46)
  Month 3 | 3.67 (0.48)
  Month 4 | 3.58 (0.72)
  Month 5 | 3.71 (0.46)
  Month 6 | 3.67 (0.48)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

41. Secondary Outcome: Parents' Perception of the Change in Child's Health Compared to One Month Ago - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 40
Time Frame: Monthly from Baseline to Month 6.
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 3.17 (0.48)
  Month 1 | 3.58 (0.72)
  Month 2 | 3.63 (0.77)
  Month 3 | 3.71 (0.86)
  Month 4 | 3.75 (0.74)
  Month 5 | 3.54 (0.72)
  Month 6 | 3.83 (0.87)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.4598, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p = 0.23, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p = 0.0806, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p = 0.0969, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p = 0.6098, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p = 0.0369, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

42. Secondary Outcome: Change in Child's Energy Levels as Reported by Parents - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 40
Time Frame: Monthly from Baseline to Month 6.
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 3.88 (0.80)
  Month 1 | 4.21 (0.66)
  Month 2 | 4.04 (0.75)
  Month 3 | 4.29 (0.69)
  Month 4 | 4.46 (0.59)
  Month 5 | 4.33 (0.64)
  Month 6 | 4.38 (0.65)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.0384, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p = 0.6328, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p = 0.0026, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p = 0.0012, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p = 0.0118, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p = 0.0221, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

43. Secondary Outcome: Changes in Limitations When Completing High-Intensity Activity - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where lower scores indicate better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the NuBest group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.13 (0.34)
  Month 1 | 1.17 (0.38)
  Month 2 | 1.21 (0.41)
  Month 3 | 1.17 (0.48)
  Month 4 | 1.08 (0.28)
  Month 5 | 1.13 (0.45)
  Month 6 | 1.04 (0.20)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

44. Secondary Outcome: Changes in Limitations When Completing Moderate-Intensity Activity - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 43
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.21 (0.41)
  Month 1 | 1.13 (0.34)
  Month 2 | 1.13 (0.34)
  Month 3 | 1.08 (0.28)
  Month 4 | 1.00 (0.00)
  Month 5 | 1.08 (0.41)
  Month 6 | 1.00 (0.00)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

45. Secondary Outcome: Changes in Limitations When Moving Around - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 43
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.00 (0.00)
  Month 1 | 1.08 (0.28)
  Month 2 | 1.08 (0.28)
  Month 3 | 1.04 (0.20)
  Month 4 | 1.00 (0.00)
  Month 5 | 1.08 (0.41)
  Month 6 | 1.00 (0.00)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

46. Secondary Outcome: Changes in Limitations When Walking 100 Meters or Climbing a Flight of Stairs - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 43
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.21 (0.66)
  Month 1 | 1.08 (0.28)
  Month 2 | 1.13 (0.34)
  Month 3 | 1.04 (0.20)
  Month 4 | 1.04 (0.20)
  Month 5 | 1.08 (0.41)
  Month 6 | 1.00 (0.00)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

47. Secondary Outcome: Changes in Limitations When Bending, Lifting, or Stooping - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 43
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.04 (0.20)
  Month 1 | 1.08 (0.28)
  Month 2 | 1.08 (0.28)
  Month 3 | 1.00 (0.00)
  Month 4 | 1.00 (0.00)
  Month 5 | 1.08 (0.41)
  Month 6 | 1.00 (0.00)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

48. Secondary Outcome: Changes in Limitations in the Kind of Schoolwork or Activities Undertaken - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 43
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.08 (0.28)
  Month 1 | 1.13 (0.34)
  Month 2 | 1.13 (0.34)
  Month 3 | 1.08 (0.28)
  Month 4 | 1.00 (0.00)
  Month 5 | 1.08 (0.41)
  Month 6 | 1.00 (0.00)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

49. Secondary Outcome: Changes in Limitations in the Amount of Time Spent Completing Schoolwork or Activities - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 43
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.13 (0.34)
  Month 1 | 1.25 (0.53)
  Month 2 | 1.08 (0.28)
  Month 3 | 1.17 (0.38)
  Month 4 | 1.00 (0.00)
  Month 5 | 1.08 (0.41)
  Month 6 | 1.00 (0.00)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

50. Secondary Outcome: Changes in Limitations During the Completion of Schoolwork or Activities - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 43
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.13 (0.34)
  Month 1 | 1.17 (0.38)
  Month 2 | 1.21 (0.66)
  Month 3 | 1.13 (0.34)
  Month 4 | 1.00 (0.00)
  Month 5 | 1.08 (0.41)
  Month 6 | 1.00 (0.00)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

51. Secondary Outcome: Change in Parents' Perception of Child's Health Compared to Other Children - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "My child seems less healthy than other children". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the NuBest group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 1.71 (0.75)
  Month 1 | 1.46 (0.59)
  Month 2 | 1.54 (0.83)
  Month 3 | 1.29 (0.46)
  Month 4 | 1.33 (0.48)
  Month 5 | 1.46 (0.51)
  Month 6 | 1.50 (0.51)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p = 0.3682, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p = 0.6098, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

52. Secondary Outcome: Change in Parents' Perception of Child's Immunity - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "When something is going around my child usually catches it". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the NuBest group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 2.38 (0.65)
  Month 1 | 2.21 (0.41)
  Month 2 | 2.00 (0.42)
  Month 3 | 2.13 (0.54)
  Month 4 | 2.13 (0.61)
  Month 5 | 2.04 (0.75)
  Month 6 | 2.08 (0.65)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p = 0.5691, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p = 0.6983, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

53. Secondary Outcome: Change in Parents' Worry About Child's Health - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "I worry more about my child's health than other parents do their children". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the NuBest group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 2.38 (0.92)
  Month 1 | 2.17 (0.70)
  Month 2 | 2.38 (0.65)
  Month 3 | 2.13 (0.68)
  Month 4 | 2.08 (0.58)
  Month 5 | 2.33 (0.82)
  Month 6 | 2.21 (0.78)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p = 0.819, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p = 0.5749, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p = 0.4873, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p = 0.9998, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p = 0.819, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

54. Secondary Outcome: Change in Parent-reported Frequency of Child's Stomach Aches - NuBest Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the NuBest group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 2.42 (0.72)
  Month 1 | 2.17 (0.48)
  Month 2 | 2.13 (0.54)
  Month 3 | 2.08 (0.65)
  Month 4 | 2.13 (0.61)
  Month 5 | 1.92 (0.50)
  Month 6 | 1.88 (0.61)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p = 0.8495, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p = 0.1951, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p = 0.0806, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis

55. Secondary Outcome: Change in Parent-reported Frequency of Child's Difficulty Going to the Toilet - NuBest Group Only (Within-Group Analysis)
Description: as for outcome 54
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale
  Baseline | 2.33 (0.92)
  Month 1 | 2.13 (0.80)
  Month 2 | 1.96 (0.62)
  Month 3 | 1.79 (0.66)
  Month 4 | 1.71 (0.62)
  Month 5 | 1.71 (0.62)
  Month 6 | 1.63 (0.58)
Statistical Analysis 1: Comparison: Intervention Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Intervention Arm; Test type: Superiority; p = 0.6983, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Intervention Arm; Test type: Superiority; p = 0.1062, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Intervention Arm; Test type: Superiority; p = 0.0333, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Intervention Arm; Test type: Superiority; p = 0.0734, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Intervention Arm; Test type: Superiority; p = 0.0219, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

56. Secondary Outcome: Changes in Overall Health as Reported by Parents - Placebo Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Parents were required to rate their child's overall health in the past four weeks. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Very Poor" ," 5 = "Excellent"). An increase in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the Placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 4.05 (0.80)
  Month 1 | 4.19 (0.87)
  Month 2 | 4.14 (0.73)
  Month 3 | 4.43 (0.68)
  Month 4 | 4.19 (0.75)
  Month 5 | 4.38 (0.59)
  Month 6 | 4.38 (0.74)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

57. Secondary Outcome: Change in Parents' Perception of the Child's Health in the Future - Placebo Group Only (Within-Group Analysis)
Description: Hide Description:
  This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Very Poor" ," 5 = "Excellent"). An increase in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 3.48 (0.60)
  Month 1 | 3.43 (0.60)
  Month 2 | 3.48 (0.75)
  Month 3 | 3.62 (0.50)
  Month 4 | 3.62 (0.50)
  Month 5 | 3.62 (0.50)
  Month 6 | 3.67 (0.58)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

58. Secondary Outcome: Parents' Perception of the Change in Child's Health Compared to One Month Ago - Placebo Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where higher scores indicate better outcomes (e.g., 1 = "Very Poor" ," 5 = "Excellent"). An increase in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 3.29 (0.72)
  Month 1 | 3.52 (0.75)
  Month 2 | 3.57 (1.08)
  Month 3 | 3.90 (0.89)
  Month 4 | 3.71 (0.90)
  Month 5 | 4.05 (0.92)
  Month 6 | 4.05 (0.97)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p = 0.982, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.091, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p = 0.4449, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p = 0.0204, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p = 0.0256, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

59. Secondary Outcome: Change in Child's Energy Levels as Reported by Parents - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 58
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 3.86 (0.73)
  Month 1 | 3.95 (0.67)
  Month 2 | 4.29 (0.64)
  Month 3 | 4.33 (0.66)
  Month 4 | 4.10 (0.70)
  Month 5 | 4.29 (0.72)
  Month 6 | 4.33 (0.66)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.9821, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p = 0.0403, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.0638, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p = 0.7195, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p = 0.1856, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p = 0.1222, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

60. Secondary Outcome: Changes in Limitations When Completing High-Intensity Activity - Placebo Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where lower scores indicate better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.38 (0.67)
  Month 1 | 1.24 (0.54)
  Month 2 | 1.24 (0.54)
  Month 3 | 1.14 (0.48)
  Month 4 | 1.14 (0.48)
  Month 5 | 1.10 (0.30)
  Month 6 | 1.19 (0.68)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

61. Secondary Outcome: Changes in Limitations When Completing Moderate-Intensity Activity - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 60
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.29 (0.56)
  Month 1 | 1.24 (0.54)
  Month 2 | 1.19 (0.51)
  Month 3 | 1.10 (0.30)
  Month 4 | 1.05 (0.22)
  Month 5 | 1.10 (0.30)
  Month 6 | 1.14 (0.48)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

62. Secondary Outcome: Changes in Limitations When Moving Around - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 60
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.10 (0.44)
  Month 1 | 1.14 (0.48)
  Month 2 | 1.10 (0.44)
  Month 3 | 1.10 (0.44)
  Month 4 | 1.14 (0.48)
  Month 5 | 1.10 (0.30)
  Month 6 | 1.19 (0.51)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

63. Secondary Outcome: Changes in Limitations When Walking 100 Meters or Climbing a Flight of Stairs - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 60
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.14 (0.36)
  Month 1 | 1.14 (0.36)
  Month 2 | 1.05 (0.22)
  Month 3 | 1.05 (0.22)
  Month 4 | 1.10 (0.30)
  Month 5 | 1.05 (0.22)
  Month 6 | 1.24 (0.62)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

64. Secondary Outcome: Changes in Limitations When Bending, Lifting, or Stooping - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 60
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.24 (0.70)
  Month 1 | 1.14 (0.36)
  Month 2 | 1.10 (0.30)
  Month 3 | 1.10 (0.30)
  Month 4 | 1.19 (0.51)
  Month 5 | 1.05 (0.22)
  Month 6 | 1.14 (0.36)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

65. Secondary Outcome: Changes in Limitations in the Kind of Schoolwork or Activities Undertaken - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 60
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.43 (0.93)
  Month 1 | 1.19 (0.51)
  Month 2 | 1.19 (0.68)
  Month 3 | 1.14 (0.48)
  Month 4 | 1.10 (0.30)
  Month 5 | 1.10 (0.30)
  Month 6 | 1.10 (0.30)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

66. Secondary Outcome: Changes in Limitations in the Amount of Time Spent Completing Schoolwork or Activities - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 60
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.43 (0.93)
  Month 1 | 1.10 (0.30)
  Month 2 | 1.19 (0.51)
  Month 3 | 1.14 (0.48)
  Month 4 | 1.14 (0.48)
  Month 5 | 1.10 (0.30)
  Month 6 | 1.10 (0.30)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

67. Secondary Outcome: Changes in Limitations During the Completion of Schoolwork or Activities - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 60
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.48 (0.87)
  Month 1 | 1.24 (0.54)
  Month 2 | 1.29 (0.64)
  Month 3 | 1.10 (0.44)
  Month 4 | 1.10 (0.30)
  Month 5 | 1.05 (0.22)
  Month 6 | 1.05 (0.22)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p = 0.982, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

68. Secondary Outcome: Change in Parents' Perception of Child's Health Compared to Other Children - Placebo Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "My child seems less healthy than other children". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the Placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.48 (0.60)
  Month 1 | 1.57 (0.75)
  Month 2 | 1.38 (0.59)
  Month 3 | 1.43 (0.60)
  Month 4 | 1.48 (0.60)
  Month 5 | 1.52 (0.75)
  Month 6 | 1.43 (0.60)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 3 vs Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 vs Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 vs Baseline; Within-group analysis only

69. Secondary Outcome: Change in Parents' Perception of Child's Immunity - Placebo Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "When something is going around my child usually catches it". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 2.24 (0.89)
  Month 1 | 2.24 (0.62)
  Month 2 | 2.19 (0.75)
  Month 3 | 2.19 (0.75)
  Month 4 | 2.14 (0.73)
  Month 5 | 2.00 (0.71)
  Month 6 | 2.05 (0.86)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p = 0.9951, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.999, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p = 0.9913, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p = 0.4517, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p = 0.8187, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

70. Secondary Outcome: Change in Parents' Worry About Child's Health - Placebo Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. The parents were asked to respond to the following statement "I worry more about my child's health than other parents do their children". Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 2.24 (0.89)
  Month 1 | 2.19 (1.03)
  Month 2 | 2.10 (1.00)
  Month 3 | 2.19 (1.03)
  Month 4 | 2.14 (1.01)
  Month 5 | 2.05 (0.80)
  Month 6 | 1.90 (1.09)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p = 0.998, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p = 0.9591, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.9994, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p = 0.9936, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p = 0.8526, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p = 0.4375, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

71. Secondary Outcome: Change in Parent-reported Frequency of Child's Stomach Aches - Placebo Group Only (Within-Group Analysis)
Description: This parameter was assessed using a parent-completed questionnaire. Responses were collected using a 5-point Likert scale with textual anchors and transformed into a numerical scale from 1 to 5, where a decrease in score indicates better outcomes (e.g., 1 = "Never," 5 = "Always"). A decrease in the mean score is associated with improvement in this parameter. This analysis summarizes the mean score at each timepoint for the placebo group only.
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 2.24 (0.77)
  Month 1 | 2.05 (0.74)
  Month 2 | 1.90 (0.70)
  Month 3 | 1.81 (0.75)
  Month 4 | 1.90 (1.00)
  Month 5 | 1.86 (0.79)
  Month 6 | 1.81 (0.68)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p = 0.7477, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.297, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p = 0.3503, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p = 0.297, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p = 0.4449, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

72. Secondary Outcome: Change in Parent-reported Frequency of Child's Difficulty Going to the Toilet - Placebo Group Only (Within-Group Analysis)
Description: as for outcome 71
Time Frame: Monthly from Baseline to Month 6
Population: Within-group analysis. No between-group comparison reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Arm
Number analyzed (Participants) | 21
score on a scale
  Baseline | 1.90 (0.94)
  Month 1 | 1.81 (0.75)
  Month 2 | 1.71 (0.72)
  Month 3 | 1.52 (0.68)
  Month 4 | 1.57 (0.68)
  Month 5 | 1.48 (0.75)
  Month 6 | 1.67 (0.73)
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 1 versus Baseline; Within-group analysis only
Statistical Analysis 2: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 2 versus Baseline; Within-group analysis only
Statistical Analysis 3: Comparison: Placebo Arm; Test type: Superiority; p = 0.9188, t-test, 2 sided — Month 3 versus Baseline; Within-group analysis only
Statistical Analysis 4: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 4 versus Baseline; Within-group analysis only
Statistical Analysis 5: Comparison: Placebo Arm; Test type: Superiority; p = 0.3503, t-test, 2 sided — Month 5 versus Baseline; Within-group analysis only
Statistical Analysis 6: Comparison: Placebo Arm; Test type: Superiority; p > 0.9999, t-test, 2 sided — Month 6 versus Baseline; Within-group analysis only

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Intervention Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT06704178/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT06704178/ICF_001.pdf